CLINICAL TRIAL: NCT06691633
Title: Postoperative Pain and Analgesic Requirements After Preoperative Methadone for Primary Total Knee Arthroplasty, a Prospective, Randomized Study
Brief Title: Postoperative Pain and Analgesic Requirements After Preoperative Methadone for Primary TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Arthur Malkani, Orthopedic Surgeon, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 23.0752
Record Dates: First submitted 2024-11-12; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: osteoarthritis; knee; total knee arthroplasty; prospective RCT; preoperative analgesia; Methadone
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Prospective, randomized cohort analysis study
Who Masked: Participant, Investigator
Masking Description: Clinical staff other than the anesthesia providers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methadone Group (Experimental): Participant receives a one-time preoperative dose of 10 mg of methadone
  Interventions: Drug: Preoperative Methadone
- Oxycodone Group (Active Comparator): participant receives a one-time preoperative dose of 10 mg of oral oxycodone
  Interventions: Drug: Preoperative Oxycodone

INTERVENTIONS:
Drug: Preoperative Methadone — patient receives a one-time preoperative dose of 10 mg of methadone
  Arms: Methadone Group
Drug: Preoperative Oxycodone — patient receives a one-time preoperative dose of 10 mg of oral oxycodone
  Arms: Oxycodone Group

SUMMARY:
The goal of this prospective, randomized study is to compare the outcomes of two cohorts of patients undergoing primary Total Knee Arthroplasty (TKA) and to determine whether a single dose of methadone administered preoperatively is effective at reducing postoperative opioid usage and postoperative pain versus a control group of patients receiving standard intraoperative opioids only for primary TKA.

The main questions it aims to answer are:

* What is the efficacy of a single preoperative dose of methadone in reducing opioid consumption and postoperative pain in primary total knee arthroplasty?
* Will the study results demonstrate the effectiveness and safety of a single preoperative dose of methadone (10 mg) in primary total knee arthroplasty in reducing postoperative opioid usage while maintaining a similar or better level of pain control when compared to a standard pain control regimen? Researchers will compare Methadone to a standard pain control regimen (Oxycodone) to see if Methadone is equivalent or more effective at reducing opioid consumption and postoperative pain in primary total knee arthroplasty

Participants will:

* be randomized into one of two groups
* undergo a primary TKA
* complete a tracking sheet documenting daily pain medicine usage and VAS pain level for the first 14 days following the TKA
* return to office at 2 weeks and 6 weeks postop for follow-up
* complete additional questionnaires at 2 weeks and 6 weeks postop

ELIGIBILITY:
Inclusion Criteria:

1. Patient age is 21-89 at time of surgery
2. Patient is scheduled to undergo a unilateral primary TKA, secondary to osteoarthritis
3. Patient agrees to participate as a study subject and signs the Informed Consent and Research Authorization document
4. Patient is able to read and speak English.

Exclusion Criteria:

1. Patient is under the age of 21
2. Patient's primary diagnosis is not osteoarthritis
3. Patient is unable to read and speak English
4. History of liver or kidney disease,
5. Known or suspected GI obstruction
6. Hypersensitivity to methadone
7. Patients with significant respiratory depression
8. Pregnant or nursing females

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Daily Opioid Use | 2 weeks
  Daily Opioid Use as measured in MME recorded daily for the first two weeks following TKA
Total opioid usage over two weeks | 2 weeks
  total daily opioid usage (as measured in MME) during the first 14 days following TKA
Visual Analogue Scale pain score | 2 weeks
  Visual Analogue Scale knee pain score (minimum value: 0, maximum value: 10). Higher scores equate to a worse outcome (a score of zero = pain free).

SECONDARY OUTCOMES:
Hospital Length of Stay | Up to 2 weeks
  Number of days patient was an inpatient in the hospital prior to discharge date
Discharge location | 2 weeks
  Whether patient was discharged to home or to a rehab facility
Two and six-week narcotic refill | 6 weeks
  Whether patient was prescribed a two week and/or six-week postoperative narcotic refill
Knee Injury and Osteoarthritis Outcome Score, Joint Replacement score | preoperatively and 6 weeks (± 2 weeks) postoperatively
  The Knee Injury and Osteoarthritis Outcome Score, Joint Replacement (KOOS, JR.) is a survey measuring overall knee health for individuals post total knee arthroplasty (TKA) by evaluating stiffness, pain, function, and activities of daily living. The minimum value is 0, the maximum value is 100. A higher score means a better outcome.
ROM | preoperatively, 2 weeks and 6 weeks (± 2 weeks) postoperatively
  active range-of-motion (ROM) as measured in degrees of extension and degrees of flexion

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Zamora, MD, Study Chair — University of Louisville
Locations (1):
- UofL Health, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
Will not share IPD if it is not a requirement

REFERENCES:
- [Background] Ferrari A, Coccia CP, Bertolini A, Sternieri E. Methadone--metabolism, pharmacokinetics and interactions. Pharmacol Res. 2004 Dec;50(6):551-9. doi: 10.1016/j.phrs.2004.05.002. PMID 15501692
- [Background] Ebert B, Thorkildsen C, Andersen S, Christrup LL, Hjeds H. Opioid analgesics as noncompetitive N-methyl-D-aspartate (NMDA) antagonists. Biochem Pharmacol. 1998 Sep 1;56(5):553-9. doi: 10.1016/s0006-2952(98)00088-4. PMID 9783723
- [Background] Duellman TJ, Gaffigan C, Milbrandt JC, Allan DG. Multi-modal, pre-emptive analgesia decreases the length of hospital stay following total joint arthroplasty. Orthopedics. 2009 Mar;32(3):167. PMID 19309064
- [Background] Davis AM, Inturrisi CE. d-Methadone blocks morphine tolerance and N-methyl-D-aspartate-induced hyperalgesia. J Pharmacol Exp Ther. 1999 May;289(2):1048-53. PMID 10215686
- [Background] Chui PT, Gin T. A double-blind randomised trial comparing postoperative analgesia after perioperative loading doses of methadone or morphine. Anaesth Intensive Care. 1992 Feb;20(1):46-51. doi: 10.1177/0310057X9202000109. PMID 1609941
- [Background] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Background] Bahreini M, Jalili M, Moradi-Lakeh M. A comparison of three self-report pain scales in adults with acute pain. J Emerg Med. 2015 Jan;48(1):10-8. doi: 10.1016/j.jemermed.2014.07.039. Epub 2014 Sep 27. PMID 25271179
- [Background] Aasvang EK, Lunn TH, Hansen TB, Kristensen PW, Solgaard S, Kehlet H. Chronic pre-operative opioid use and acute pain after fast-track total knee arthroplasty. Acta Anaesthesiol Scand. 2016 Apr;60(4):529-36. doi: 10.1111/aas.12667. Epub 2015 Dec 28. PMID 26708043